CLINICAL TRIAL: NCT01536990
Title: Sensitivity to Change of the Lower Extremity Functional Scale and a Single-Item Functional Assessment Tool in Patients With Neurological Impairments Secondary to Stroke
Brief Title: Sensitivity to Change of the Lower Extremity Functional Scale in Patients With Stroke
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 06-002770
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Lower Extremity Dysfunction; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stroke: Medically stable patients receiving inpatient or outpatient physical therapy care for lower extremity dysfunction secondary to stroke.

SUMMARY:
The purpose of this study was to investigate the reliability, construct validity, and sensitivity to change of the Lower Extremity Functional Scale (LEFS) in individuals affected by stroke.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the reliability, construct validity, and sensitivity to change of the Lower Extremity Functional Scale (LEFS) in individuals affected by stroke. Patients were measured with the LEFS at the beginning and end of physical therapy treatment, or at 8 weeks of physical therapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable patients receiving inpatient or outpatient physical therapy care for lower extremity dysfunction due to stroke

Exclusion Criteria:

* Unable to understand English
* More than moderate assist for bed mobility and coming to sitting from the supine position
* Lower extremity amputation
* Unable to reach overhead, grasp an object, or feed self with an upper extremity

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medically stable patients receiving inpatient or outpatient physical therapy care for lower extremity dysfunction due to stroke.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
LEFS | 36 days average (range 4-76 days)
  Lower Extremity Function Scale

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Verheijde, PhD MBA PT, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States